CLINICAL TRIAL: NCT00935077
Title: A Collaborative Model to Improve BP Control and Minimize Racial Disparities-CCC
Brief Title: A Collaborative Model to Improve Blood Pressure (BP) Control and Minimize Racial Disparities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01HL091841 (NIH)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension; Asthma
Keywords: Hypertension; Pharmacist Physician Collaborative Management of Hypertension
MeSH Terms: conditions — Hypertension; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 24 Month PPCM BP (Experimental): A 24 month long physician/pharmacist collaborative intervention is implemented to manage hypertension
  Interventions: Other: 24 Month PPCM BP
- 9 Month PPCM BP (Experimental): A 9 month long physician/pharmacist collaborative intervention is implemented to manage hypertension
  Interventions: Other: 9 Month PPCM BP
- PPCM Asthma (Sham Comparator): A 9 month long physician/pharmacist collaborative intervention is implemented to manage asthma
  Interventions: Other: PPCM Asthma
- BP Control Arm (No Intervention): No PPCM intervention

INTERVENTIONS:
Other: PPCM Asthma — Pharmacists collaborate with physicians to manage asthma
  Arms: PPCM Asthma
Other: 24 Month PPCM BP — Pharmacists collaborate with physicians for 24 months to manage hypertension.
  Arms: 24 Month PPCM BP
Other: 9 Month PPCM BP — Pharmacists collaborate with pharmacists for 9 months to manage hypertension
  Arms: 9 Month PPCM BP

SUMMARY:
The purpose of the study is to determine the degree to which pharmacist-physician collaborative management (PPCM) of hypertension can be adopted and implemented in clinics with geographic and racial diversity and whether patients in clinics which implement PPCM achieve greater blood pressure control than patients in clinics which do not implement PPCM.

Primary Hypothesis: BP control at 9 months will be significantly greater in patients from clinics randomized to the two PPCM BP intervention groups compared to the control group.

DETAILED DESCRIPTION:
Blood pressure (BP) is controlled in only 34% of patients with high BP, leading to unnecessary strokes, myocardial infarctions and other cardiovascular events. BP control can be improved with physician/ pharmacist collaborative management (PPCM). Our long-range goal is to achieve excellent BP control rates using PPCM that can be implemented in private practices in diverse communities. The objective of this application is to conduct a large multi-center clinical trial in clinics with geographic, racial and ethnic diversity to determine the extent to which the model is implemented. This practice-based research network (PBRN) is unique with a large minority population and great diversity in operation and community size. This prospective, cluster-randomized trial uses 27 clinics, matched and randomized to the active intervention (2 groups) or a control group in 648 patients. Following 9 months of the intervention, one intervention group will continue the intervention following 9 months while the other will discontinue it. We will also randomize 18 patients per clinic into a passive observation group (n=486) to determine if PPCM is implemented more broadly in the clinic. Patients in all three groups will be followed for 24 months. We will accomplish our objectives and test our central hypothesis by pursing the following aims:

Aim 1: To determine if patients in clinics randomized to PPCM can achieve better BP control at 9 months compared to patients in clinics randomized to the control group.

Primary Hypothesis: BP control at 9 months will be significantly greater in patients from clinics randomized to the two PPCM BP intervention groups compared to the control group.

Aim 2: To determine if patients in clinics randomized to continuation of PPCM achieve better long-term BP control compared to patients in clinics randomized to discontinuation of PPCM after 9 months and to patients in control clinics.

Our innovative approach addresses critical organizational barriers and challenges existing approaches to achieving better BP control. This study is novel because it will: 1) be the largest study to test this model, 2) use a cluster randomized design to include many more clinics than previously used, 3) use a diverse group of clinics with broad geographic distribution, 4) include large numbers of patients from minority groups to assess potential health disparities, 5) evaluate whether the effect can be sustained long-term, 6) include standardized BP measurements rather than error-prone office BPs, 7) minimize selection bias, and 8) evaluate a "passive observation group" to evaluate dissemination of PPCM throughout the practice. We expect that our study will find a 6-8 mm Hg difference in systolic BP which would lead to 20-30% fewer coronary deaths and 25-40% fewer stroke deaths if applied across broadly across similar settings.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish speaking males or females, over 18 years of age with a diagnosis of hypertension,
2. have uncontrolled BP defined as > 140 mm Hg SBP or > 90 mm Hg DBP for patients with uncomplicated hypertension; or > 130 mm Hg SBP or > 80 mm Hg DBP for patients with diabetes or chronic kidney disease, and
3. receive care from one of the participating clinics.

Exclusion Criteria:

1. current signs of hypertensive emergency (acute angina, stroke, or renal failure;
2. severe HTN (systolic BP >200 or diastolic BP > 114 mm Hg);
3. history of MI, stroke, or unstable angina in the prior 6 months;
4. systolic dysfunction with a LV ejection fraction < 35% documented by echocardiography, nuclear medicine study, or ventriculography;
5. renal insufficiency, defined by a glomerular filtration rate less than 20 ml/min or previously documented proteinuria > 1 gram per day;
6. significant hepatic disease, including prior diagnoses of cirrhosis, Hepatitis B or C infection, or laboratory abnormalities (serum ALT or AST > 2 times control or total bilirubin > 1.5 mg/dl) in the prior 6 months;
7. pregnancy;
8. diagnoses of pulmonary hypertension or sleep apnea (unless treated by continuous positive pressure ventilation);
9. poor prognosis with a life expectancy estimated less than 2 years;
10. residence in a nursing home or diagnosis of dementia; and
11. inability to give informed consent or impaired cognitive function (defined as > 3 errors on the 10-item Pfeiffer Portable Mental Status Questionnaire, administered during study intake).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1441 (Actual)
Dates: Start 2010-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control | 9 Months

SECONDARY OUTCOMES:
Blood Pressure Control | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Carter, PharmD, Principal Investigator — University of Iowa
Locations (28):
- United States (28):
  - University of California San Diego, San Diego, California
  - St. Francis Hospital Medical Center, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Idaho State University, Pocatello, Idaho
  - Midwestern University, Downers Grove, Illinois
  - Genesis Health System, Davenport, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - The University of Iowa, Iowa City, Iowa
  - Siouxland Medical Education Foundation, Sioux City, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - SUNY-University of Buffalo, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Regional Health Service District, Spartanburg, South Carolina
  - Texas Tech University Health Science Center, Amarillo, Texas
  - Seton Healthcare, Austin, Texas
  - University of Texas at El Paso, El Paso, Texas
  - Memorial Hermann Hospital System, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
  - Wheaton Franciscan Medical Group, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Anderegg MD, Gums TH, Uribe L, MacLaughlin EJ, Hoehns J, Bazaldua OV, Ives TJ, Hahn DL, Coffey CS, Carter BL. Pharmacist Intervention for Blood Pressure Control in Patients with Diabetes and/or Chronic Kidney Disease. Pharmacotherapy. 2018 Mar;38(3):309-318. doi: 10.1002/phar.2083. Epub 2018 Feb 23. PMID 29331037
- [Derived] Anderegg MD, Gums TH, Uribe L, Coffey CS, James PA, Carter BL. Physician-Pharmacist Collaborative Management: Narrowing the Socioeconomic Blood Pressure Gap. Hypertension. 2016 Nov;68(5):1314-1320. doi: 10.1161/HYPERTENSIONAHA.116.08043. Epub 2016 Sep 6. PMID 27600181
- [Derived] Carter BL. Primary Care Physician-Pharmacist Collaborative Care Model: Strategies for Implementation. Pharmacotherapy. 2016 Apr;36(4):363-73. doi: 10.1002/phar.1732. Epub 2016 Apr 6. PMID 26931738
- [Derived] Isetts BJ, Buffington DE, Carter BL, Smith M, Polgreen LA, James PA. Evaluation of Pharmacists' Work in a Physician-Pharmacist Collaborative Model for the Management of Hypertension. Pharmacotherapy. 2016 Apr;36(4):374-84. doi: 10.1002/phar.1727. Epub 2016 Mar 18. PMID 26893135
- [Derived] Carter BL, Coffey CS, Ardery G, Uribe L, Ecklund D, James P, Egan B, Vander Weg M, Chrischilles E, Vaughn T. Cluster-randomized trial of a physician/pharmacist collaborative model to improve blood pressure control. Circ Cardiovasc Qual Outcomes. 2015 May;8(3):235-43. doi: 10.1161/CIRCOUTCOMES.114.001283. Epub 2015 Mar 24. PMID 25805647
- [Derived] Carter BL, Coffey CS, Uribe L, James PA, Egan BM, Ardery G, Chrischilles EA, Ecklund D, Vander Weg M, Vaughn T; Collaboration Among Pharmacists and Physicians to Improve Outcomes Now (CAPTION) trial investigators. Similar blood pressure values across racial and economic groups: baseline data from a group randomized clinical trial. J Clin Hypertens (Greenwich). 2013 Jun;15(6):404-12. doi: 10.1111/jch.12091. Epub 2013 Apr 1. PMID 23730989
- [Derived] Demik DE, Vander Weg MW, Lundt ES, Coffey CS, Ardery G, Carter BL. Using theory to predict implementation of a physician-pharmacist collaborative intervention within a practice-based research network. Res Social Adm Pharm. 2013 Nov-Dec;9(6):719-30. doi: 10.1016/j.sapharm.2013.01.003. Epub 2013 Mar 16. PMID 23506651
- [Derived] Carter BL, Clarke W, Ardery G, Weber CA, James PA, Vander Weg M, Chrischilles EA, Vaughn T, Egan BM; Collaboration Among Pharmacists Physicians To Improve Outcomes Now (CAPTION) Trial Investigators. A cluster-randomized effectiveness trial of a physician-pharmacist collaborative model to improve blood pressure control. Circ Cardiovasc Qual Outcomes. 2010 Jul;3(4):418-23. doi: 10.1161/CIRCOUTCOMES.109.908038. PMID 20647575